CLINICAL TRIAL: NCT04450446
Title: Restart Anticoagulation in Patients With Spontaneous Intracerebral Hemorrhage and Mechanical Heart Valves
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-315
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cerebral hemorrhage
  Interventions: Drug: Low molecular weight heparin
- thromboembolism
  Interventions: Drug: Low molecular weight heparin
- no thromboembolism and cerebral hemorrhage
  Interventions: Drug: Low molecular weight heparin

INTERVENTIONS:
Drug: Low molecular weight heparin — Anticoagulation therapy

SUMMARY:
The investigators retrospectively reviewed the electronic medical records of the patients with spontaneous cerebral hemorrhage and mechanical valves from 2015 to 2020 in the second affiliated hospital of Zhejiang university medical college. Medical documents and patient data were reviewed, including patient age, gender, type of mechanical heart valve, replacement time, replacement site, underlying disease, anticoagulant drugs at admission, type of cerebral hemorrhage, treatment mode, time without anticoagulant, length of stay, mortality, etc

ELIGIBILITY:
Inclusion Criteria:

* patients with spontaneous cerebral hemorrhage and mechanical valves

Exclusion Criteria:

* age<18y
* pregnant patients
* death in 24 hours without anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with spontaneous cerebral hemorrhage and mechanical valves from 2015 to 2020 in the second affiliated hospital of Zhejiang university medical college.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
survival and death patients after follow-up investigation for 60 months | 2015-2020
  the patients with spontaneous cerebral hemorrhage and mechanical valves in the second affiliated hospital of Zhejiang university medical college.

CONTACTS AND LOCATIONS:
Overall Officials: libin li, MD, Study Director — second affiliated hospital,school of medicine, zhejiang university,china
Locations (2):
- China (2):
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang
  - Second Affiliated Hospital,School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No